CLINICAL TRIAL: NCT04375696
Title: Randomized Double Blind Placebo Controlled Clinical Study to Evaluate the Effect on Weight of a Medical Device With Polyglucosamine L 112 in a Group of Overweight and Obese Subjects: POSO Study (Polyglucosamine and Overweight)
Brief Title: Randomized Double Blind Placebo Controlled Clinical Trial to Evaluate Obese and Overweight Subjects
Acronym: POSO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Certmedica International GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IT-1501202
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Weight Loss
Keywords: Polyglucosamine; Formoline L112; Medical Device
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Product (Experimental): 75 subjects of both sexes suffering from overweight and mild obesity BMI 25-32 and weigh in > 75 kg
  Interventions: Drug: Polyglucosamine L112
- Placebo (Placebo Comparator): 75 subjects of both sexes suffering from overweight and mild obesity BMI 25-32 and weigh in > 75 kg
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Polyglucosamine L112 — Polyglucosamine; Ascorbic Acid; Tartaric Acid
  Other Names: Formoline L112
  Arms: Product
Other: Placebo — Dicalcium Phosphate; Microcrystalline Cellulose; Iron Oxide (yellow, brown, and black); Magnesium Stearate; Silicon Dioxide
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the effect on weight loss in a group of subjects suffering from overweight and mild obesity (BMI between 25 and 32 Kg/m2) and with weight > 75 Kg/m2 being administered with a 3 g/day polyglucosamine dosage.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the effect on weight loss in a group of subjects suffering from overweight and mild obesity (BMI between 25 and 32 Kg/m2) and with weight > 75 Kg/m2 being administered with a 3 g/day polyglucosamine dosage.

The secondary objectives of the study are:

* to evaluate the effect of supplementation on blood triglyceride levels
* to evaluate the effect of supplementation on blood levels of Total Cholesterol (CT), LDL, and HDL
* to evaluate the effect of supplementation on glucose, insulin, insulin resistance assessed by calculating the Homeostatic metabolic assessment (HOMA)
* to evaluate the effect of supplementation on liver enzymes (transaminases) and renal function (creatinine)
* to evaluate the effect of supplementation on BMI (Body Mass Index)
* to evaluate the effect of supplementation on the abdominal circumference
* to evaluate the effect of supplementation on body composition evaluated by dual X-ray densitometer (DXA)
* to evaluate the effect of supplementation on the serum levels of reactive oxygen species
* to evaluate the effect of supplementation on serum antioxidant capacity

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age between 18-65
* Both sexes - mandatory adequate contraceptive method for women in fertility age
* BMI between 25-32 kg/m2 and weigh in > 75 kg, with no previous diet-therapy attempts with at least a 5% weight loss in the last year
* No 3 kg weight fluctuation in the last 3 months
* Beck Depression Inventory (BDI) score < 20
* Binge Eating Scale (BES) score < 27

Exclusion Criteria:

* Shellfish allergy or to any other ingredient in the product
* Previous diet-therapy attempts with at least a 5% weight loss in the last year
* 3 kg weight fluctuation in the last 3 months
* Presumed or confirmed pregnancy
* No contraceptive method for women in fertility age
* Cardiopathies, nephropathies, hepatopathies, bronchopneumopathies, hemopathies dermopathies clinically significant chronic degenerative CNS (Central Nervous System) diseases
* Active peptic ulcer, ulcerative colitis, Crohn disease, celiac disease, inflammatory bowel disease
* Alcoholism
* Epilepsy
* Past or current malignancies
* Intellectual disability
* Significant motor disability
* Drug abuse
* Autoimmune diseases
* Symptomatic cholelithiasis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 3-month treatment
  To evaluate the weight loss with 3 g/die administration of polyglucosamine (PG)

SECONDARY OUTCOMES:
Triglycerides | 3-month treatment
  To evaluate the effect of PG administration on triglycerides plasma levels
Cholesterol | 3-month treatment
  To evaluate the effect of PG administration on total cholesterol plasma levels
HOMA | 3-month treatment
  To evaluate the effect of PG administration on glucose, insulin, insulin resistance (measured through Homeostatic Metabolic Assessment - HOMA
Hepatic Enzymes - Renal Functionality | 3-month treatment
  To evaluate the effect of PG administration on transaminases and creatinine
BMI | 3-month treatment
  To evaluate the effect of PG administration on BMI
Abdominal Circumference | 3-month treatment
  To evaluate the effect of PG administration on the abdominal circumference
DXA | 3-month treatment
  To evaluate the effect of PG administration on corporeal composition by means of DXA (Dual energy X-ray Absorptiometry)
ROS | 3-month treatment
  To evaluate the effect of PG administration on ROS (Reactive Oxygen Species) serum levels
Antioxidant Serum Capacity | 3-month treatment
  To evaluate the effect of PG administration on serum antioxidant capacity

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Rondanelli, Prof., Principal Investigator — University of Pavia
Locations (1):
- Azienda di Servizi alla Persona Istituzioni Assistenziali Riunite di Pavia, Pavia, Lombardy, Italy

REFERENCES:
- [Derived] Rondanelli M, Perna S, Porta MD, Lombardoni F, Patelli Z, Nichetti M, Gasparri C, Pistolesi E, Cestaro B, Cazzola R. Modification of metabolic syndrome parameters following the administration of polyglucosamine L112: results of a subgroup analysis of subjects enrolled in a double blind randomised placebo controlled clinical investigation. BMC Nutr. 2025 Sep 2;11(1):170. doi: 10.1186/s40795-025-01153-8. PMID 40898346